CLINICAL TRIAL: NCT04159636
Title: Comparison of the Risk of Pulmonary Aspiration Assessed by Gastric Ultrasound in Elderly Patients in Fasting Group vs. Carbohydrate Loading Group
Brief Title: Pulmonary Aspiration in Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Eunah Cho, MD, Clinical Assistant Professor, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KBSMC 2019-10-013
Record Dates: First submitted 2019-11-03; First posted 2019-11-12 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting group (No Intervention): Participants will be remained fasted until surgery
- Carbohydrate group (Experimental): Participants will be allowed to drink carbohydrate beverage before 2 hours of surgery
  Interventions: Other: Carbohydrate beverage

INTERVENTIONS:
Other: Carbohydrate beverage — The participants in this group are allowed to drink carbohydrate until 2 hours before surgery
  Arms: Carbohydrate group

SUMMARY:
The aim of this study was to compare the risk of pulmonary aspiration assessed with gastric ultrasonography in elderly patients, undergoing elective surgery.

DETAILED DESCRIPTION:
Recently, carbohydrate loading is suggested for enhanced recovery after surgery.

Aging process often accompanies gastrointestinal dysmotility. Therefore, elderly patients might have undiagnosed gastro-esophageal reflux disease, or other gastrointestinal disorders. Moreover, because of their co-morbid underlying diseases and multi-drug effects, gastric emptying might be further delayed in the elderly patients.

This study was designated to compared the risk of pulmonary aspiration in elderly patients, with gastric ultrasound between fasting group and carbohydrate loading group.

ELIGIBILITY:
Inclusion Criteria:

* aged from 65
* scheduled for elective surgery
* American Society of Anesthesiologists physical status 1 or 2

Exclusion Criteria:

* Diagnosed for diseases that might delay gastric emptying (obesity, diabetes, hiatal hernia, gastro-esophageal reflux disease, ileus)
* psychiatric or mental disorders
* delirium
* dementia
* parkinsonism
* alcoholism
* drug abuse

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2020-08-06 (Actual); Study Completion 2020-08-06 (Actual)

PRIMARY OUTCOMES:
Incidence of risk of pulmonary aspiration assessed by gastric ultrasound defined by Perlas grade 2 | 2 hours after intake of last allowable carbohydrate drink time
  Incidence of Perlas grade 2. Clear fluid is detected in gastric antrum by gastric antral ultrasound on both supine and right lateral decubitus position.
  Perlas grade 2: fluid appears in both supine and right lateral decubitus positions Perlas grade 1: fluid is detected only in right decubitus position Perlas grade 0: fluid is not detected in both supine and right lateral decubitus positions.

SECONDARY OUTCOMES:
cross-sectional area of gastric antrum in supine position | 2 hours after intake of last allowable carbohydrate drink time
  cross sectional area of gastric antrum is calculated by using the following formula: cross-sectional area = long axis x short axis x 3.14 /4
cross-sectional area of gastric antrum in right decubitus position | 2 hours after intake of last allowable carbohydrate drink time
  cross sectional area of gastric antrum is calculated by using the following formula: cross-sectional area = long axis x short axis x 3.14 /4

CONTACTS AND LOCATIONS:
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea